CLINICAL TRIAL: NCT07278206
Title: Mitigating Cognitive Problems and Fatigue With Brain Stimulation in Long COVID
Brief Title: Brain Stimulation in Long COVID
Acronym: MALIBU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Post Covid Netwerk Nederland (Unknown)
Responsible Party: Principal Investigator, Sander Verfaillie, Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL-009207; 11080022420018 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-11-19; First posted 2025-12-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Long COVID; PASC Post Acute Sequelae of COVID 19; Post COVID-19 Condition (PCC)
Keywords: TMS; PASC; long COVID; PCC; neuroimaging; non-invasive brain stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and the investigators conducting neuropsychological assessment and doing data analysis will remain blinded to treatment allocation. Due to the nature of the intervention, rTMS technicians cannot be blinded. However, they will be asked not to reveal allocation to participants and other researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Experimental): The active intervention will consist of high-frequency rTMS delivered to the left dorsolateral prefrontal cortex (DLPFC). Stimulation will be administered at 10 Hz frequency, 110% of the individual's resting motor threshold and then adjusted for the individual cortex-skull distance, with 3,000 pulses per session with a total duration of 30 minutes (60 trains of 5 seconds, 25-second inter-train intervals).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham-stimulation will be administered at 60% motor threshold at the same location (left DLPFC) using a placebo coil, which is identical to the stimulation coil in appearance, but with a built-in metal plate that blocks most of the active stimulation while maintaining mechanical scalp sensation.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The active intervention will consist of high-frequency (10 Hz) TMS delivered to the left dorsolateral prefrontal cortex (DLPFC), at 110% of the individual's resting motor threshold, adjusted for the individual cortex-skull distance, with 3,000 pulses per session with a total duration of 30 minutes (60 trains of 5 seconds, 25-second inter-train intervals). Sham-stimulation will be administered at 60% motor threshold at the same location (left DLPFC) using a placebo coil, which is identical to the stimulation coil in appearance, but with a built-in metal plate that blocks most of the active stimulation while maintaining mechanical scalp sensation. The stimulation target will be individualized using functional MRI data acquired during a Tower of London planning task allowing neuronavigation to the site of task-related activation. Each participant will receive four sessions per week for six weeks, totaling 24 sessions.
  Other Names: rTMS; TMS; non-invasive brain stimulation; NIBS
  Arms: Active rTMS
Device: Sham device — Sham-stimulation will be administered at 60% motor threshold at the left DLPFC using a placebo coil, which is identical to the stimulation coil in appearance, but with a built-in metal plate that blocks most of the active stimulation while maintaining mechanical scalp sensation. 3,000 pulses per session will be applied with a total duration of 30 minutes (60 trains of 5 seconds, 25-second inter-train intervals). The stimulation target will be individualized using functional MRI data acquired during a Tower of London planning task, allowing neuronavigation to the site of task-related activation. Each participant will receive four sessions per week for six weeks, totaling 24 sessions.
  Other Names: Sham rTMS; Sham TMS; Placebo; Placebo coil
  Arms: Sham rTMS

SUMMARY:
Cognitive problems and severe fatigue are two frequently occurring symptoms in long COVID, also known as Post-Covid Condition or Post-Acute Sequelae of COVID-19 (PASC), and their causes are currently unknown. Previous studies have shown reduced blood flow and increased inflammation in the brains of people with PASC. These brain processes are related to fatigue and cognitive problems. In other conditions, these disrupted brain processes have been treated safely and successfully with non-invasive brain stimulation. This may offer an effective treatment for people with PASC.

The main goal of this clinical trial is to see whether non-invasive brain stimulation called repetitive transcranial magnetic stimulation (rTMS) can reduce fatigue in adults with PASC who also have trouble concentrating. rTMS uses short magnetic pulses on the scalp to gently stimulate a small brain area.

In this study, 66 adults with PASC will be included, recruited through the Post-COVID Network Netherlands. Participants will be randomly assigned to receive either active rTMS or sham (placebo) rTMS. Sham rTMS feels and looks similar to the active treatment, but it does not generate effective magnetic pulses. The brain area that will be targeted is personalized using a brain scan (MRI) during a planning task. All participants will receive 24 rTMS sessions over six weeks (four per week).

Fatigue will be measured within two weeks before and two weeks after treatment to determine whether active rTMS works better than sham. We will also look at cognition, brain connectivity and blood flow, signs of (neuro)inflammation, daily activity using an activity watch, and questionnaires about quality of life, mood, and sleep. Follow-up on cognition and questionnaires will take place 3 and 6 months after the end of the treatment.

DETAILED DESCRIPTION:
Background Long COVID, also known as Post-COVID Condition (PCC) or Post-Acute Sequelae of COVID-19 (PASC), is characterized by persistent symptoms following SARS-CoV-2 infection without an alternative explanation. Fatigue and cognitive dysfunction are among the most common and disabling complaints, with substantial effects on daily functioning, work participation, and quality of life. Converging evidence from neuroimaging and fluid biomarkers points to altered cerebral perfusion, disrupted functional connectivity, and neuroinflammatory processes in at least a subset of people with PASC.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technique that can modulate cortical excitability and large-scale networks, with downstream effects on cerebral blood flow, connectivity and inflammatory signaling. Small, uncontrolled studies in PASC and related fatigue conditions suggest potential benefits of rTMS for fatigue and cognition, but placebo-controlled evidence in PASC is lacking and prior studies have used relatively few sessions. The present trial addresses this gap by testing a functional magnetic resonance (fMRI)-guided rTMS protocol in a randomized, double-blind design, while characterizing neurobiological mechanisms of change.

Objectives The primary objective is to determine whether high-frequency (10 Hz) rTMS reduces fatigue severity in adults with PASC compared with sham stimulation. Secondary objectives are to evaluate effects on physical and cognitive functioning, patient-reported outcome measures (e.g., mood, sleep, and quality of life), to quantify rTMS-related changes in neuroimaging and blood-based biomarkers reflecting neuronal integrity, cerebral perfusion, and (neuro)inflammation, and to examine whether these biomarkers can predict symptom improvement.

Design and procedures This is a single-center, randomized, double-blind, sham-controlled clinical trial. Sixty-six adults with PASC characterized by severe fatigue and cognitive complaints will be enrolled through the Post-COVID Network Netherlands. After baseline assessments, participants are randomized 1:1 to active rTMS or sham rTMS using block randomization implemented in Castor EDC with allocation concealment; participants and outcome assessors are blinded.

Treatment is delivered four times per week for six consecutive weeks (24 sessions). A minimum effective dose of 16 sessions applies when burden needs to be reduced. Outcome assessments are conducted within two weeks before the treatment at baseline (T0), within two weeks after the intervention period (T1), and at follow-up three months (T2) and six months (T3) after treatment to evaluate long-term effects. During the six-week intervention period a brief subset of patient-reported measures is collected weekly to monitor symptom trajectories and adverse effects.

Neuroimaging and blood sampling are obtained at T0 and T1. The MRI protocol (3T Siemens VIDA) includes structural, perfusion (ASL), resting-state and task-based fMRI (Tower of London), spectroscopy (MRS), and conventional FLAIR/SWI. Blood-derived biomarkers (e.g., NfL, GFAP, brain-derived tau, IL-6/IL-1/TNF-α, CCL11, BDNF) are assayed from EDTA plasma with standardized handling and storage prior to batch analysis. Actigraphy is assessed over 8 days prior to treatment and 8 days following treatment, and heart-rate variability is assessed during 4 nights and 4 times directly after waking for 5 minutes 2 weeks before treatment and directly after treatment.

Interventions Active treatment consists of high-frequency (10 Hz) rTMS delivered to the left dorsolateral prefrontal cortex at 110% resting motor threshold, with intensity adjusted for scalp-to-cortex distance. The stimulation target is individualized using task-based fMRI activation from a Tower of London planning task and neuronavigation (Localite). Sham sessions are performed with a placebo coil, that mimics sound and sensation, and at 60% motor threshold, so that it delivers no effective magnetic field. Participants and researchers involved in clinical assessments, data collection, and analysis remain blinded to allocation; technicians are trained to avoid any disclosure that could compromise masking. To enhance feasibility for participants with fatigue and sensory sensitivity, the treatment environment is kept low-stimulus with reduced lighting and noise, scheduling is flexible with a weekly buffer option, and the minimum 16-session option supports completion.

Endpoints and analysis The primary endpoint is change in fatigue from baseline to post-treatment, analyzed as the between-group difference in pre- to post-treatment change under the intention-to-treat principle. Secondary endpoints span cognitive functioning, mood, sleep, quality of life, and physical performance, together with multimodal neuroimaging and blood-based biomarkers that analyse neuronal integrity, cerebral blood flow, functional connectivity, and inflammation. Statistical analyses use linear mixed-effects models with appropriate covariates and multiplicity is handled via Bonferroni for secondary endpoints and FDR for neuroimaging and exploratory analyses.

Safety and ethics Safety is monitored throughout treatment and follow-up via standardized AE questionnaires and weekly tolerability questions. Known contraindications to rTMS/MRI are applied at screening, and procedures for managing common side effects and rare events are in place. The study is conducted per the Declaration of Helsinki and national regulations, with approval by the METc Amsterdam UMC. Participants provide written informed consent, travel costs are reimbursed, and a small participation compensation is provided.

Recruitment and setting Recruitment is coordinated through the Post Covid Network Netherlands patient portal, enabling efficient identification of potentially eligible individuals who consented to be approached for research. The trial is conducted at Amsterdam UMC.

Conclusion If the intervention proves effective, this study will provide the first placebo-controlled evidence for high-frequency rTMS to reduce fatigue in long COVID, with neuroimaging and blood biomarkers to shed light on underlying disease and treatment mechanisms. Even if no between-group difference is observed, the trial will yield valuable information on PASC and underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Meet the World Health Organization (WHO) definition of long COVID.
* Aged 18 years or older.
* Severe fatigue, defined as a score ≥35 on the Checklist Individual Strength (CIS) fatigue subscale.
* Significant cognitive complaints, defined as a score ≥18 on the CIS concentration subscale.
* Commitment to actively undergo rTMS
* Ability to attend the study site regularly for treatment sessions.
* Capacity to provide written informed consent.

Exclusion Criteria:

* Prior rTMS treatment or current intensive/experimental treatment for long COVID.
* History of epilepsy or first-degree family history of epilepsy.
* Recent initiation or dosage change of psychotropic medication (less than six weeks for psychotropic medication including antidepressants and antipsychotic drugs, less than two weeks for benzodiazepines). Medication doses must remain stable during the study.
* Other active concurrent pharmacological treatments for post-covid symptoms
* Contraindications to MRI scanning (e.g., non-removable metallic implants, severe claustrophobia).
* Presence of a cochlear implant.
* Neurological disorders such as multiple sclerosis or other neurodegenerative conditions.
* Pregnancy.
* Known brain lesions or ischaemic scars influencing seizure threshold.
* Severe uncontrolled migraines.
* Severe cardiovascular disease
* Raised intracranial pressure.
* High alcohol consumption (males/females: 21/14 units per week) or use of epileptogenic drugs.
* Severe sleep deprivation at the time of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-11-17 (Estimated); Study Completion 2029-05-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Fatigue will be measured within two weeks before and within two weeks after treatment, and at 3 and 6 months follow-up.
  Fatigue as measured by the 8-item fatigue subscale of the Checklist Individual Strength (CIS). The subscale is scored on a 7-point Likert scale, adding up to a total score between 8 and 56. A score of 35 or higher indicates the presence of severe fatigue.

SECONDARY OUTCOMES:
Objective cognitive functioning | Objective cognitive functioning will be measured two weeks before and two weeks after treatment and at 3 and 6 months follow-up after treatment.
  Objective cognitive functioning will be measured using a composite score that combines the T-scores from multiple cognitive tests: (1) Stroop Test (information processing and interference sensitivity), (2) Trail Making Test A/B (various domains of executive function), (3) D2 Test (selective and sustained attention, concentration, and processing speed), and (4) 15-Word Test (memory).
  These scores will be combined into a composite score by taking the mean of the individual T-scores, which are corrected for age, sex, and education and will provide a comprehensive assessment of objective cognitive functioning. The final composite score will not include any individual test units but will provide an overall score reflecting performance across multiple cognitive domains.
Arterial Spin Labeling (ASL) | Neuroimaging will be performed within two weeks before and within two weeks after treatment.
  We will measure blood-brain barrier integrity and perfusion using ASL.
Magnetic Resonance Spectroscopy (MRS) | Neuroimaging will be performed within two weeks before and within two weeks after treatment.
  Neuroinflammation and neuronal injury will be measured using MRS (metabolites for inflammation include choline, creatine and myo-inositol, and for neuronal injury N-acetyl-aspartate, glutamate and lactate).
Functional Magnetic Resonance Imaging (fMRI) | Neuroimaging will be performed within two weeks before and within two weeks after treatment.
  Participants will undergo a 10-minute resting-state scan, during which they are instructed to relax and remain awake while looking at a visual fixation cross for the entirety of the scan. After the resting-state scan, participants will complete the Tower of London task to measure task-based activity.
Actigraphy | Continuous period of eight days two weeks before and directly after treatment
  Participants will wear an Actiwatch to monitor actigraphy for a continuous period of five days. Participants will be instructed to wear the actiwatch continuously during the measurement days and to maintain their usual daily routines. Actigraphy data will provide objective measures of day and nighttime activity.
Short physical performance battery (SPPB) | Physical performance will be measured within two weeks before and within two weeks after treatment and at three and six months after treatment (follow-up).
  The short physical performance battery (SPPB) will be performed to measure physical performance through three components: gait speed, balance, and repeated chair stands. The SPPB score is a composite of three physical tasks (gait speed, balance, and repeated chair stands) combined into a single score, ranging from 0-12. Higher scores mean better physical performance.
Simple Reaction Time (SRT) | Participants will complete the SRT within two weeks before, within two weeks after treatment and three and six months after treatment (follow-up).
  Reaction time will be assessed using a Simple Reaction Time (SRT) task, where participants are instructed to press the spacebar as quickly as possible when red circles appears on the screen. The task consists of 25 trials, with a randomized interval between each trial. The primary outcome will be the mean reaction time, with secondary analysis of the coefficient of variation (CV) across trials.
Effort-based decision task | The effort-based decision task will be completed within two weeks before and within two weeks after treatment.
  An effort-based decision task will be assessed to measure reward sensitivity. In this task, participants will either accept or reject offers in which they could exert physical effort (ticking boxes on screen, 5 levels) to gain rewards (money, 5 levels).
Neurofilament light (NF-L) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Neurofilament light (NF-L) will be quantified to reflect neuronal injury.
Brain-Derived Tau (BD-Tau) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Brain-Derived Tau (BD-Tau) will be quantified to reflect neuronal injury.
Interleukin-6 (IL-6) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis.Interleukin-6 (IL-6) will be quantified to measure (neuro)inflammation.
Interleukin-1 (IL-1) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Interleukin-1 (IL-1) will be quantified to measure (neuro)inflammation.
Glial Fibrillary Acidic Protein (GFAP) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Glial Fibrillary Acidic Protein (GFAP) will be quantified to measure astrocytic activity
Tumor Necrosis Factor-alpha (TNF-α) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Tumor Necrosis Factor-alpha (TNF-α) will be quantified to measure (neuro)inflammation.
Eotaxin-1/CCL11 | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Eotaxin-1/CCL11 will be quantified to measure (neuro)inflammation.
Brain-derived neurotrophic factor (BDNF) | Blood samples will be collected within two weeks before and within two weeks after treatment.
  Blood will be drawn from the antecubital vein into EDTA tubes, placed on ice, centrifuged, and plasma stored at -80°C until analysis. Brain-derived neurotrophic factor (BDNF) will be quantified as a brain plasticity marker.
Checklist Individuele Spankracht (CIS) | Survey will be completed within two weeks before and within two weeks after treatment, and three and six months after treatment (follow-up).
  The Checklist Individuele Spankracht (CIS) measures subjective fatigue and related behavior. Score ranges from 20-140, with higher scores indicating worse outcomes.
Cognitive Failures Questionnaire (CFQ) | Survey will be completed within two weeks before and within two weeks after treatment, and three and six months after treatment (follow-up).
  The Cognitive Failures Questionnaire (CFQ) measures subjective cognition. Score ranges from 0-100, with higher scores indicating worse outcomes (greater cognitive failures).
Illness Perception Questionnaire (IPQ)-short form | Survey will be completed within two weeks before and within two weeks after treatment.
  The Illness Perception Questionnaire (IPQ)-short form assesses various dimensions of an individual's illness perception, including its perceived consequences, timeline, controllability, and emotional representation. The responses to each question are evaluated individually, as no composite score is generated. Higher scores on each question indicate worse perceptions.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Survey will be completed within two weeks before treatment, weekly during treatment and within two weeks after treatment.
  The PROMIS-29 will measure a multi-domain scale that measures physical function, fatigue, pain interference, anxiety, depression, sleep disturbance, and ability to participate in social roles. The PROMIS-Cognitive function 8a will assess subjective cognitive function.
  For most PROMIS instruments, a score of 50 represents the average for the general U.S. population, with a standard deviation of 10. Higher T-scores reflect more of the concept being measured (e.g., higher cognitive function). For example, a T-score of 60 is one standard deviation above average (better than average) and a T-score of 40 is one standard deviation below average (worse than average).
Patient Health Questionnaire 9 (PHQ-9) | Survey will be completed within two weeks before treatment, weekly during treatment, within two weeks after treatment and at three and six months after treatment (follow-up).
  The Patient Health Questionnaire 9 (PHQ-9) measures the severity of depressive symptoms, including mood and sleep. The score ranges from 0 to 27, with higher scores indicating worse outcomes. It includes a question specifically about suicidality (Item 9), which will be used to monitor thoughts of self-harm or suicide throughout the study.
DePaul Symptom Questionnaire (DSQ)- post-exterional malaise and postural orthostatic tachycardia syndrome related questions | Survey will be completed within two weeks before treatment, within two weeks after treatment and at three and six months after treatment (follow-up).
  Using the DePaul Symptom Questionnaire (DSQ) the severity of symptoms related to post-exertional malaise and postural orthostatic tachycardia syndrome will be assessed. Higher scores indicate worse outcomes (more severe symptoms).
Bell Chronic Fatigue Syndrome Disability Scale | Survey will be completed within two weeks before treatment, within two weeks after treatment and at three and six months after treatment (follow-up).
  The Bell chronic fatigue syndrome disability scale consists of one question that measures the degree of disability, focusing on the impact of the illness on daily functioning. A higher score means a greater degree of disability.
Insomnia Severity Index (ISI) | Survey will be completed within two weeks before treatment, within two weeks after treatment and at three and six months after treatment (follow-up).
  The insomnia severity index (ISI) evaluates the severity of insomnia symptoms, including difficulty falling asleep, staying asleep, and daytime impairment due to sleep problems. The score ranges from 0 to 28, with higher scores indicating worse outcomes.
Jacobson Fatigue Catastrophizing Scale (J-FCS) | Survey will be completed within two weeks before treatment and within two weeks after treatment.
  The Jacobson Fatigue Catastrophizing Scale (J-FCS) assesses how individuals catastrophize or worry about their fatigue, including thoughts and feelings that amplify the experience of fatigue. The score ranges from 10 to 50, with higher scores indicating a higher degree of catastrophic thinking.
Self-Efficacy Scale 28 (SES-28) | Survey will be completed within two weeks before treatment and within two weeks after treatment.
  The Self-Efficacy Scale 28 (SES-28) consists of a 7-item questionnaire measuring self-efficacy and coping of difficult or stressful situations. The score ranges from 7 to 28, with higher scores reflecting a higher degree of self-efficacy.
Cognitive and Behavioral Responses to Symptoms Questionnaire (CBRQ) | Survey will be completed within two weeks before treatment and within two weeks after treatment.
  The Cognitive and Behavioral Responses to Symptoms Questionnaire (CBRQ) 16-item questionnaire is used to assess fear avoidance, damage beliefs, and all-or-nothing behavior. Items are scored on a 5-point scale, with higher scores indicating a stronger presence of the specific cognitive or behavioral response.
Treatment Inventory of Costs in Patients (TIC-P) - Work Absenteeism/Productivity Subscale | Survey will be completed within two weeks before treatment and at three and six months after treatment (follow-up).
  The Treatment Inventory of Costs in Patients (TIC-P) - Work Absenteeism/Productivity Subscale assesses the impact of illness on work attendance and productivity. It does not provide a single score but instead measures whether the individual is currently working, whether they are required to stay home from work due to their condition, and how many days of work are missed due to illness. This information helps evaluate the effect of illness on work performance and productivity.
Multimodal Evaluation of Sensory Sensitivity (MESSY) - multisensory, visual and auditory sensitivity subscales | Survey will be completed within two weeks before treatment, within two weeks after treatment and three and six months after treatment (follow-up).
  The Multimodal Evaluation of Sensory Sensitivity (MESSY) - multisensory, visual and auditory sensitivity subscales assess sensory sensitivity across these three sensory modalities. Every item is measured on a 1 to 5 point scale. A higher score indicates a higher sensory sensitivity severity.
Credibility Expectancy Questionnaire (CEQ) | Survey will be completed within two weeks before treatment.
  The Credibility Expectancy Questionnaire (CEQ) assesses the credibility and expectations of patients regarding the intervention, measuring how much they believe in its potential effectiveness. It consists of three questions regarding credibility and three questions regarding expectancy, each question rated or converted to a 9 point Likert scale. A higher score means higher treatment credibility and expectancy.

OTHER OUTCOMES:
Heart rate variability (HRV) | Four nights and four mornings two weeks before and directly after treatment
  Participation in HRV measurements is voluntary, and data will be collected only from participants who consent to this component. The Polar H10 will be worn during sleep and for 5 minutes immediately upon waking each day to capture nocturnal and early-morning HRV metrics. HRV will provide indices of autonomic nervous system function.

CONTACTS AND LOCATIONS:
Overall Officials: Sander C.J. Verfaillie, Dr., Principal Investigator — Amsterdam UMC, GGZ InGeest; Odile A van den Heuvel, Prof. Dr., Study Chair — Amsterdam UMC; Ysbrand D van der Werf, Prof. Dr., Study Chair — Amsterdam UMC; Esmée Verwijk, Dr., Study Chair — University of Amsterdam, Amsterdam UMC; Céline N Dietz, MSc/MA, Study Director — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zingaropoli MA, Pasculli P, Barbato C, Petrella C, Fiore M, Dominelli F, Latronico T, Ciccone F, Antonacci M, Liuzzi GM, Talarico G, Bruno G, Galardo G, Pugliese F, Lichtner M, Mastroianni CM, Minni A, Ciardi MR. Biomarkers of Neurological Damage: From Acute Stage to Post-Acute Sequelae of COVID-19. Cells. 2023 Sep 13;12(18):2270. doi: 10.3390/cells12182270. PMID 37759493
- [Background] Yang G, Gu R, Kubo J, Kakuda W. Is the efficacy of repetitive transcranial magnetic stimulation influenced by baseline severity of fatigue symptom in patients with myalgic encephalomyelitis. Int J Neurosci. 2020 Jan;130(1):64-70. doi: 10.1080/00207454.2019.1663189. Epub 2019 Sep 13. PMID 31483181
- [Background] Verveen A, Verfaillie SCJ, Visser D, Koch DW, Verwijk E, Geurtsen GJ, Roor J, Appelman B, Boellaard R, van Heugten CM, Horn J, Hulst HE, de Jong MD, Kuut TA, van der Maaden T, van Os YMG, Prins M, Visser-Meily JMA, van Vugt M, van den Wijngaard CC, Nieuwkerk PT, van Berckel B, Tolboom N, Knoop H. Neuropsychological functioning after COVID-19: Minor differences between individuals with and without persistent complaints after SARS-CoV-2 infection. Clin Neuropsychol. 2025 Feb;39(2):347-362. doi: 10.1080/13854046.2024.2379508. Epub 2024 Jul 17. PMID 39016843
- [Background] Verveen A, Verfaillie SCJ, Visser D, Csorba I, Coomans EM, Koch DW, Appelman B, Barkhof F, Boellaard R, de Bree G, van de Giessen EM, Golla S, van Heugten CM, Horn J, Hulst HE, de Jong MD, Kuut TA, van der Maaden T, van Os YMG, Prins M, Slooter AJC, Visser-Meily JMA, van Vugt M, van den Wijngaard CC, Nieuwkerk PT, Knoop H, Tolboom N, van Berckel BNM. Neurobiological basis and risk factors of persistent fatigue and concentration problems after COVID-19: study protocol for a prospective case-control study (VeCosCO). BMJ Open. 2023 Jun 30;13(6):e072611. doi: 10.1136/bmjopen-2023-072611. PMID 37399444
- [Background] van den Heuvel OA, Van Gorsel HC, Veltman DJ, Van Der Werf YD. Impairment of executive performance after transcranial magnetic modulation of the left dorsal frontal-striatal circuit. Hum Brain Mapp. 2013 Feb;34(2):347-55. doi: 10.1002/hbm.21443. Epub 2011 Nov 11. PMID 22076808
- [Background] Thaweethai, T., Jolley, S. E., Karlson, E. W., Levitan, E. B., Levy, B., McComsey, G. A., McCorkell, L., Nadkarni, G. N., Parthasarathy, S., Singh, U., Walker, T. A., Selvaggi, C. A., Shinnick, D. J., Schulte, C. C. M., Atchley-Challenner, R., Horwitz, L. I., Foulkes, A. S., Alba, G. A., Alicic, R., … Zisis, S. (2023). Development of a Definition of Postacute Sequelae of SARS-CoV-2 Infection. JAMA, 329(22). https://doi.org/10.1001/jama.2023.8823
- [Background] Schultheiss C, Willscher E, Paschold L, Gottschick C, Klee B, Henkes SS, Bosurgi L, Dutzmann J, Sedding D, Frese T, Girndt M, Holl JI, Gekle M, Mikolajczyk R, Binder M. The IL-1beta, IL-6, and TNF cytokine triad is associated with post-acute sequelae of COVID-19. Cell Rep Med. 2022 Jun 21;3(6):100663. doi: 10.1016/j.xcrm.2022.100663. PMID 35732153
- [Background] Scholing JM, Lambregts BIHM, van den Bosch R, Aarts E, van der Schaaf ME. Greater fatigue is more strongly associated with reduced reward sensitivity in the long-term phase of coronavirus disease (COVID-19) than in the early phase. Brain Behav Immun Health. 2025 Jul 5;48:101056. doi: 10.1016/j.bbih.2025.101056. eCollection 2025 Oct. PMID 40686929
- [Background] Sasaki N, Yamatoku M, Tsuchida T, Sato H, Yamaguchi K. Effect of Repetitive Transcranial Magnetic Stimulation on Long Coronavirus Disease 2019 with Fatigue and Cognitive Dysfunction. Prog Rehabil Med. 2023 Feb 28;8:20230004. doi: 10.2490/prm.20230004. eCollection 2023. PMID 36861061
- [Background] Santana K, Franca E, Sato J, Silva A, Queiroz M, de Farias J, Rodrigues D, Souza I, Ribeiro V, Caparelli-Daquer E, Teixeira AL, Charvet L, Datta A, Bikson M, Andrade S. Non-invasive brain stimulation for fatigue in post-acute sequelae of SARS-CoV-2 (PASC). Brain Stimul. 2023 Jan-Feb;16(1):100-107. doi: 10.1016/j.brs.2023.01.1672. Epub 2023 Jan 21. PMID 36693536
- [Background] Sack AT, Cohen Kadosh R, Schuhmann T, Moerel M, Walsh V, Goebel R. Optimizing functional accuracy of TMS in cognitive studies: a comparison of methods. J Cogn Neurosci. 2009 Feb;21(2):207-21. doi: 10.1162/jocn.2009.21126. PMID 18823235
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Reggente N, Moody TD, Morfini F, Sheen C, Rissman J, O'Neill J, Feusner JD. Multivariate resting-state functional connectivity predicts response to cognitive behavioral therapy in obsessive-compulsive disorder. Proc Natl Acad Sci U S A. 2018 Feb 27;115(9):2222-2227. doi: 10.1073/pnas.1716686115. Epub 2018 Feb 12. PMID 29440404
- [Background] Peljto AL, Barker-Cummings C, Vasoli VM, Leibson CL, Hauser WA, Buchhalter JR, Ottman R. Familial risk of epilepsy: a population-based study. Brain. 2014 Mar;137(Pt 3):795-805. doi: 10.1093/brain/awt368. Epub 2014 Jan 26. PMID 24468822
- [Background] Pagliaccio D, Middleton R, Hezel D, Steinman S, Snorrason I, Gershkovich M, Campeas R, Pinto A, Van Meter P, Simpson HB, Marsh R. Task-based fMRI predicts response and remission to exposure therapy in obsessive-compulsive disorder. Proc Natl Acad Sci U S A. 2019 Oct 8;116(41):20346-20353. doi: 10.1073/pnas.1909199116. Epub 2019 Sep 23. PMID 31548396
- [Background] Oostra E, Jazdzyk P, Vis V, Dalhuisen I, Hoogendoorn AW, Planting CHM, van Eijndhoven PF, van der Werf YD, van den Heuvel OA, van Exel E. More rTMS pulses or more sessions? The impact on treatment outcome for treatment resistant depression. Acta Psychiatr Scand. 2025 Apr;151(4):485-505. doi: 10.1111/acps.13768. Epub 2024 Nov 21. PMID 39569643
- [Background] Nilsson J, Ekblom O, Ekblom M, Lebedev A, Tarassova O, Moberg M, Lovden M. Acute increases in brain-derived neurotrophic factor in plasma following physical exercise relates to subsequent learning in older adults. Sci Rep. 2020 Mar 10;10(1):4395. doi: 10.1038/s41598-020-60124-0. PMID 32157099
- [Background] Lind A, Boraxbekk CJ, Petersen ET, Paulson OB, Andersen O, Siebner HR, Marsman A. Do glia provide the link between low-grade systemic inflammation and normal cognitive ageing? A 1 H magnetic resonance spectroscopy study at 7 tesla. J Neurochem. 2021 Oct;159(1):185-196. doi: 10.1111/jnc.15456. Epub 2021 Jul 14. PMID 34142382
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Khullar D, Zhang Y, Zang C, Xu Z, Wang F, Weiner MG, Carton TW, Rothman RL, Block JP, Kaushal R. Racial/Ethnic Disparities in Post-acute Sequelae of SARS-CoV-2 Infection in New York: an EHR-Based Cohort Study from the RECOVER Program. J Gen Intern Med. 2023 Apr;38(5):1127-1136. doi: 10.1007/s11606-022-07997-1. Epub 2023 Feb 16. PMID 36795327
- [Background] Gelauff JM, Rosmalen JGM, Gardien J, Stone J, Tijssen MAJ. Shared demographics and comorbidities in different functional motor disorders. Parkinsonism Relat Disord. 2020 Jan;70:1-6. doi: 10.1016/j.parkreldis.2019.11.018. Epub 2019 Nov 23. PMID 31785442
- [Background] Fernandez-Castaneda A, Lu P, Geraghty AC, Song E, Lee MH, Wood J, O'Dea MR, Dutton S, Shamardani K, Nwangwu K, Mancusi R, Yalcin B, Taylor KR, Acosta-Alvarez L, Malacon K, Keough MB, Ni L, Woo PJ, Contreras-Esquivel D, Toland AMS, Gehlhausen JR, Klein J, Takahashi T, Silva J, Israelow B, Lucas C, Mao T, Pena-Hernandez MA, Tabachnikova A, Homer RJ, Tabacof L, Tosto-Mancuso J, Breyman E, Kontorovich A, McCarthy D, Quezado M, Vogel H, Hefti MM, Perl DP, Liddelow S, Folkerth R, Putrino D, Nath A, Iwasaki A, Monje M. Mild respiratory COVID can cause multi-lineage neural cell and myelin dysregulation. Cell. 2022 Jul 7;185(14):2452-2468.e16. doi: 10.1016/j.cell.2022.06.008. Epub 2022 Jun 13. PMID 35768006
- [Background] Donse L, Sack AT, Fitzgerald PB, Arns M. Sleep disturbances in obsessive-compulsive disorder: Association with non-response to repetitive transcranial magnetic stimulation (rTMS). J Anxiety Disord. 2017 Jun;49:31-39. doi: 10.1016/j.janxdis.2017.03.006. Epub 2017 Mar 31. PMID 28388457
- [Background] Caulfield KA, Fleischmann HH, Cox CE, Wolf JP, George MS, McTeague LM. Neuronavigation maximizes accuracy and precision in TMS positioning: Evidence from 11,230 distance, angle, and electric field modeling measurements. Brain Stimul. 2022 Sep-Oct;15(5):1192-1205. doi: 10.1016/j.brs.2022.08.013. Epub 2022 Aug 27. PMID 36031059
- [Background] Boissoneault J, Letzen J, Lai S, O'Shea A, Craggs J, Robinson ME, Staud R. Abnormal resting state functional connectivity in patients with chronic fatigue syndrome: an arterial spin-labeling fMRI study. Magn Reson Imaging. 2016 May;34(4):603-8. doi: 10.1016/j.mri.2015.12.008. Epub 2015 Dec 18. PMID 26708036
- [Background] Biswal B, Kunwar P, Natelson BH. Cerebral blood flow is reduced in chronic fatigue syndrome as assessed by arterial spin labeling. J Neurol Sci. 2011 Feb 15;301(1-2):9-11. doi: 10.1016/j.jns.2010.11.018. Epub 2010 Dec 16. PMID 21167506
- [Background] Ballouz T, Menges D, Anagnostopoulos A, Domenghino A, Aschmann HE, Frei A, Fehr JS, Puhan MA. Recovery and symptom trajectories up to two years after SARS-CoV-2 infection: population based, longitudinal cohort study. BMJ. 2023 May 31;381:e074425. doi: 10.1136/bmj-2022-074425. PMID 37257891
- [Background] Bai YW, Yang QH, Chen PJ, Wang XQ. Repetitive transcranial magnetic stimulation regulates neuroinflammation in neuropathic pain. Front Immunol. 2023 Apr 25;14:1172293. doi: 10.3389/fimmu.2023.1172293. eCollection 2023. PMID 37180127
- [Background] Ajcevic M, Iscra K, Furlanis G, Michelutti M, Miladinovic A, Buoite Stella A, Ukmar M, Cova MA, Accardo A, Manganotti P. Cerebral hypoperfusion in post-COVID-19 cognitively impaired subjects revealed by arterial spin labeling MRI. Sci Rep. 2023 Apr 10;13(1):5808. doi: 10.1038/s41598-023-32275-3. PMID 37037833
- [Background] Aftanas LI, Gevorgyan MM, Zhanaeva SY, Dzemidovich SS, Kulikova KI, Al'perina EL, Danilenko KV, Idova GV. Therapeutic Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Neuroinflammation and Neuroplasticity in Patients with Parkinson's Disease: a Placebo-Controlled Study. Bull Exp Biol Med. 2018 Jun;165(2):195-199. doi: 10.1007/s10517-018-4128-4. Epub 2018 Jun 19. PMID 29923005
- See also: Study website — http://www.hersenstimulatie-longcovid.nl